CLINICAL TRIAL: NCT02037958
Title: The Laryngeal Mask Airway Supreme (TM) is an Effective Alternative to Laryngoscope-guided Tracheal Intubation for Patients Undergoing Elective Laparoscopic Cholecystectomy-- A Prospective Randomized Controlled Trial
Brief Title: Laryngeal Mask Airway Supreme Versus the Tracheal Tube as an Airway Device in Elective Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Kelvin Quek How Yow, Consultant Anaesthetist, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CGHLMAS2010
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Cholecystitis; Choledocholithiasis
MeSH Terms: conditions — Cholecystitis; Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngeal Mask Airway-Supreme (Experimental): Patients who are randomly assigned to receive the LMA-Supreme
  Interventions: Device: Laryngeal Mask Airway-Supreme
- Endotracheal Tube (Active Comparator): Patients who are randomly assigned to receive endotracheal intubation
  Interventions: Device: Endotracheal Tube

INTERVENTIONS:
Device: Laryngeal Mask Airway-Supreme — Patients who receive the LMA-S
  Other Names: LMA-S; LMA-Supreme; LMA Supreme
  Arms: Laryngeal Mask Airway-Supreme
Device: Endotracheal Tube — Patients who receive endotracheal intubation
  Other Names: ETT; Tracheal Tube
  Arms: Endotracheal Tube

SUMMARY:
We hypothesise that the use of the LMA-Supreme provides greater ease of insertion and reduced haemodynamic variability during insertion compared to the tracheal tube, whilst still maintaining a patent airway to facilitate elective laparoscopic cholecystectomy in selected patients.

DETAILED DESCRIPTION:
The Laryngeal Mask Airway Supreme(LMA-S) has been used successfully to maintain a patent airway for laparoscopic surgery. Our study compares the use of LMA-S with that of the tracheal tube (ETT) with respect to the ease of insertion and potential haemodynamic disturbance during insertion.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 1 and 2
* Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* BMI > 30
* Known gastro-oesophageal reflux disease
* predicted or documented difficult airway
* contraindications to drugs in the standardized anaesthesia protocol

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time to Effective Airway | Baseline
  Time to achieve effective airway was defined as time between removing the face-mask, inserting the airway device and obtaining a sustained square-wave capnograph trace with manual ventilation

SECONDARY OUTCOMES:
Number of attempts taken for successful placement of airway device | Baseline
  Number of attempts needed for successful placement of either the LMA-Supreme or the tracheal tube, as assigned
Number of attempts taken for successful placement of gastric tube | Baseline
  Number of attempts needed for successful placement of gastric tube. Correct gastric tube placement was determined by positive suctioning of gastric contents or detection of injected air with epigastric auscultation.
Haemodynamic response to insertion of airway device | Baseline, 1 min, 5 min
  Systolic blood pressure and heart rate at 0 min, 1 min, 5 min, starting from the time the face mask was removed from the patient's face.
Peak airway pressure during pneumoperitoneum | Assessed intra-operatively, during the period of pneumoperitoneum
  Peak airway pressure recorded during pneumoperitoneum, measured during the surgery
Incidence of post-operative sore throat | Assessed 1 hr after the surgery, at the Recovery Area
  Patients were asked about the presence of sore throat - defined as the presence of constant pain in the throat, independent of swallowing, 1 hr after the end of surgery. No further follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Quek, MMED (Anaes), Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore